CLINICAL TRIAL: NCT00227981
Title: Maintenance Psychotherapies in Recurrent Depression: Study II
Brief Title: Maintenance Interpersonal Psychotherapy for Sustaining Remission of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH049115 (NIH); DSIR 950309-9905
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Depression Relapse; Maintenance Therapy
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy; Fluoxetine

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy
Drug: Fluoxetine

SUMMARY:
This study will evaluate the effectiveness of maintenance interpersonal psychotherapy (IPT) in preventing relapse of depression in women who have required combined psychotherapy and pharmacotherapy treatment to obtain a remission of depression symptoms.

DETAILED DESCRIPTION:
Depression is a serious medical illness that can recur more than once in a person's lifetime. Effective treatment methods are needed to maintain a state of remission in people who have had prior episodes of depression. IPT is a brief and highly structured type of psychotherapy that addresses interpersonal issues associated with depression. Previous studies have shown that it is an effective method for treating depression. This study will evaluate the effectiveness of maintenance ITP in preventing relapse of depression in women who have required combined psychotherapy and pharmacotherapy treatment to obtain remission of depressive symptoms.

Participants in this open label study will be recruited from a previous study, "Maintenance Psychotherapy in Recurrent Depression: Study I." In this study participants will initially receive weekly sessions of IPT as well as medication treatment with fluoxetine. Any participants who do not reach remission of depressive symptoms after 6 weeks will be given other standard treatments for depression. Once remission of depressive symptoms is reached, participants will continue receiving weekly IPT and fluoxetine treatment for 20 weeks. After 20 weeks, fluoxetine treatment will be discontinued, and all participants will receive IPT alone for 6 weeks before entering the maintenance phase of the study. Upon entrance into this phase, participants will be randomly assigned to receive IPT weekly, biweekly, or monthly for 18 months. Functioning and depressive symptoms will be assessed at Month 24.

ELIGIBILITY:
Inclusion Criteria:

* Met all entry criteria for the parent study, "Maintenance Psychotherapy in Recurrent Depression, Study I"
* Began IPT as outlined in the parent study
* Demostrated compliance with IPT sessions during the parent study
* Exhibits less than a 50% reduction in score on the Hamilton Rating Scale for Depression after 12 weeks of psychotherapy or fails to meet stabilization criteria after 24 weeks of psychotherapy during the parent study

Exclusion Criteria:

* Any unstable medical illness

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93
Dates: Start 1995-03; Study Completion 2001-03

PRIMARY OUTCOMES:
Score on the Hamilton Rating Scale for Depression (measured at Month 24)

SECONDARY OUTCOMES:
Score on the Beck Depression Inventory
Score on the Global Assessment of Functioning (measured at Month 24)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Dombrovski AY, Cyranowski JM, Mulsant BH, Houck PR, Buysse DJ, Andreescu C, Thase ME, Mallinger AG, Frank E. Which symptoms predict recurrence of depression in women treated with maintenance interpersonal psychotherapy? Depress Anxiety. 2008;25(12):1060-6. doi: 10.1002/da.20467. PMID 18781665
- [Derived] Frank E, Kupfer DJ, Buysse DJ, Swartz HA, Pilkonis PA, Houck PR, Rucci P, Novick DM, Grochocinski VJ, Stapf DM. Randomized trial of weekly, twice-monthly, and monthly interpersonal psychotherapy as maintenance treatment for women with recurrent depression. Am J Psychiatry. 2007 May;164(5):761-7. doi: 10.1176/ajp.2007.164.5.761. PMID 17475735